CLINICAL TRIAL: NCT04904510
Title: Evaluation of the INDICAID™ COVID-19 Rapid Antigen Test in Symptomatic Populations and Asymptomatic Community Testing
Brief Title: Evaluation of the INDICAID™ COVID-19 Rapid Antigen Test
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Noah Kojima, MD, Principal Investigator, University of California, Los Angeles
Other Study IDs: Pro00047510
Record Dates: First submitted 2021-05-19; First posted 2021-05-27 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Sample Collection: People routinely testing for COVID-19 would have an extra sample collected to assess the diagnostic device.
  Interventions: Diagnostic Test: INDICAID™ COVID-19 Rapid Antigen Test

INTERVENTIONS:
Diagnostic Test: INDICAID™ COVID-19 Rapid Antigen Test — The diagnostic assay will be compared to a EUA SARS-CoV-2 assay

SUMMARY:
The INDICAID™ Rapid Antigen Test was used in real-world outbreak testing. The antigen test was used together with PCR testing. This study was designed to evaluate whether the addition of a rapid antigen test decreased time to results in a real-world setting.

DETAILED DESCRIPTION:
Description of the INDICAID™ COVID-19 Rapid Antigen Test The INDICAID™ Rapid Test by PHASE Scientific is a LFA designed for the qualitative detection of SARS-CoV-2 nucleocapsid protein in nasal swab samples.

Sample collection and procedure To collect a sample, a nasal swab sample is collected by inserting the provided swab 1 inch into the nasal cavity. The swab is rubbed against the inside walls of both nostrils 5 times in a large circular path. The swab is then dipped into a buffer solution to elute the sample. Finally, three drops of the buffer solution-specimen mix are applied to the LFA test device. After 20 minutes, the user observes the test device for the presence or absence of a test line that indicates detection of the SARS-CoV-2 antigen. An Internal Quality Control line is included to indicate whether the test has been performed correctly.

COVID-19 outbreak screening with the LFA In this Dual-Track testing approach, the LFA is used to identify preliminary positives to trigger prioritization of sample processing for subsequent RT-PCR confirmatory testing.

In Approach A, a preliminary positive result from the LFA would expedite the corresponding patient VTM sample for laboratory-based RT-PCR. Expedited testing would obtain results. In Approach B, a preliminary positive result from the LFA result would trigger the testing of the corresponding patient VTM sample with an onsite rapid nucleic acid amplification test (cobas® SARS-CoV-2 & Influenza A/B Nucleic acid test on the cobas® Liat system, Roche Molecular Diagnostics). In addition to the onsite rapid RT-PCR test, the corresponding patient VTM sample was also sent for expedited laboratory-based RT-PCR testing. All samples testing negative with the LFA were sent for RT-PCR testing.

ELIGIBILITY:
Inclusion Criteria:

* at least 5 years of age and report onset
* at least two of the following COVID-19 symptoms within 5 days or less: fever or chills, fatigue, sore throat, congestion or runny nose, cough, headache, diarrhea, shortness of breath or difficulty breathing, muscle or body aches, new loss of taste or smell, nausea, or vomiting.

Exclusion Criteria:

* That do not fit inclusion criteria or vulnerable populations

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People testing for COVID at multiple sites in California
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CityHealth Urgent Care Oakland, Oakland, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Cohort: Participants were recruited from people testing for SARS-CoV-2. Those that met eligibility criteria were recruited. Among those willing to partake in the study, sample specimens were collected to assess the diagnostic device. Those results were compared to an EUA SARS-CoV-2 assay.
Period: Overall Study
Arm/Group | Study Cohort
Started | 297
Completed | 297
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Evaluation of the INDICAID™ COVID-19 Rapid Antigen Test: Sample specimens were collected from participants testing for SARS-CoV-2. Results from the diagnostic test were compared to the EUA SARS-CoV-2 assay.
Arm/Group | Evaluation of the INDICAID™ COVID-19 Rapid Antigen Test
Number analyzed (Participants) | 297
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [23 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158
  Male | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 231
  Not Hispanic or Latino | 66
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 259
  More than one race | 4
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 297

OUTCOME MEASURES:

1. Primary Outcome: Test Concordance
Description: The concordance with the INDICAID COVID-19 Rapid Antigen Test with an EUA PCR test
Time Frame: Day 1
Measure: Number (95% Confidence Interval); unit: positive percent agreement
Arm/Group | Sample Collection
Number analyzed (Participants) | 349
positive percent agreement | 85.3 [75.6 to 91.6]

ADVERSE EVENTS:
Time Frame: Participants were actively monitored on the day of the study. Participants could report adverse events to a call line after the study and the call line was monitored for 3 months.
Description: There were no adverse events.
Arm/Group | Sample Collection
All-Cause Mortality (participants affected / at risk) | 0/297
Serious Adverse Events (participants affected / at risk) | 0/297
Other Adverse Events (participants affected / at risk) | 0/297

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT04904510/Prot_SAP_000.pdf